CLINICAL TRIAL: NCT04425915
Title: Efficacy of Convalescent Plasma Therapy in Patients With COVID-19: A Randomized Control Trial
Brief Title: Efficacy of Convalescent Plasma Therapy in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-COVID-04
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-06

CONDITIONS: COVID
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma with Standard of Care (Experimental): Two doses of 250 ml Convalescent plasma from recovered COVID-19 patients + Standard of Care will be given to severely sick COVID-19 patients in the treatment arm
  Interventions: Biological: Convalescent Plasma; Other: Standard of Care
- Standard of Care (Active Comparator): The Ministry of Health and Family Welfare has issued detailed guidelines for the management of sCOVID-19 based on varying grades of severity which may be periodically updated. For the management of ARDS or sepsis the respective guidelines issued by ARDSNet and Surviving Sepsis campaign will be followed. Other institutional protocols for supportive management will be implemented. (Ref: Guidelines on Clinical Management of COVID-19. MoHFW, GoI.2020.)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Convalescent Plasma — Dose-250 ml Frequency - 2 doses on consecutive days Duration -Start by day 3 of symptom onset (of severe COVID-19 as in inclusion criteria) in eligible patients
  Arms: Convalescent Plasma with Standard of Care
Other: Standard of Care — The Ministry of Health and Family Welfare has issued detailed guidelines for the management of sCOVID-19 based on varying grades of severity which may be periodically updated. For the management of ARDS or sepsis the respective guidelines issued by ARDSNet and Surviving Sepsis campaign will be followed. Other institutional protocols for supportive management will be implemented. (Ref: Guidelines on Clinical Management of COVID-19. MoHFW, GoI.2020.)

SUMMARY:
Currently, no effective treatments are available for the COVID-19. Scientists and Researchers are working on many aspects of treatment options for the development of vaccination and medication to combat this life-threatening problem. Convalescent plasma from recovered COVID-19 patients contains antibodies against COVID-19 which may be beneficial to severely sick COVID-19 patients. Investigator have recently concluded a pilot phase II open-label RCT on the efficacy of convalescent plasma in severe COVID 19 patients in which encouraging results were seen. Investigator plan to further study the efficacy and safety of convalescent plasma in COVID-19 severely sick patients through an RCT. Investigator will collect up to 500 ml Convalescent Plasma from the COVID-19 recovered persons after 14 days of clinical recovery with two consecutive SARS CoV-2 negative tests by PCR at least 24 hours apart. This plasma will be tested and frozen and stored. On requisition it will be thawed and sent to the treating center. Two doses of 250 ml convalescent plasma each will be transfused on two consecutive days to patients who fit the eligibility criteria (Severely sick COVID-19 patients) and are randomized to the convalescent plasma group along with the standard of care and the other group will receive standard of care alone. Data will be collected to study the benefits and adverse events related to convalescent plasma transfusion.

DETAILED DESCRIPTION:
Study Centres:

Institute of Liver and Biliary Sciences Sector D-1, Vasant Kunj New Delhi -110070

- Collection and testing of Convalescent Plasma

Treatment Centres

Lok Nayak Jai Prakash Hospital (LNJP)

Rajiv Gandhi Super-speciality Hospital (RGSSH)

Methodology Donor Plasmapheresis COVID-19 recovered patients will be counseled and informed regarding convalescent plasma donation. The contact information of those who agree will be sent to the coordinator at ILBS Blood Centre.

* The prospective donor will be contacted and if willing to come for donation, the donor will be provided conveyance if required, to come to ILBS Blood centre for Plasma Donation
* At ILBS the donor will be counseled and the doctor in-charge will explain the procedure to the Donor.
* The donor will be given a Donor Information Sheet and Informed consent will be taken on the document
* The eligibility for plasma donation will be ascertained through Medical History, Physical Examination, and laboratory tests.

Donor Eligibility for Plasmapheresis

* Virologically documented (PCR positive by nasopharyngeal swab) who is recovered and free of symptoms for 14 days.
* Has tested negative for SARS CoV 2 on two consecutive tests 24 hrs apart.
* Fulfill all criteria of donor eligibility for donor Plasmapheresis under the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020
* Females who have been pregnant may be tested for anti-HLA antibodies and eligible if negative for the same.

The following Donors will be excluded

* Do not fulfill all criteria of donor eligibility for donor Plasmapheresis under
* the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020
* Females who have been pregnant and have not been tested for HLA antibodies or are HLA antibody positive if tested and previously transfused donors (to prevent TRALI)
* Donors who have taken steroids during treatment for COVID-19 Donor Selection Process
* A detailed medical history of the donor will be taken and documented
* Physical examination ( Height, Weight, Blood Pressure, Temperature, adequate veins for phlebotomy)
* Laboratory Testing: complete Blood count, Testing for hepatitis B virus, hepatitis C virus, HIV, malaria, and syphilis) by serology, blood grouping, and antibody screening. Serum protein will be done in repeat donors ( Ref: D&C Act and Rules)
* Serum COVID-19 specific IgG antibody positive (with an IgG titre higher than 80).
* All Results Evaluated & Clinically Correlated The donor is deemed eligible/non-eligible

Plasmapheresis Procedure

* Determine Volume to be collect-approx. 500 ml
* As per the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020
* Start Donor Plasmapheresis Procedure(As per SOP)
* Collect Convalescent Plasma The convalescent plasma will be properly labeled and frozen at -80o C in a separate Deep Freezer. It will not be issued to other patients who are with non-COVID.
* Label Details: As per the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020.
* Storage condition- Below -30oC
* Shelf life: - 1 Year

Other Sources of Convalescent Plasma:

Convalescent Plasma collected during a CP donation drive by Delhi Govt. following all rules and regulations of the Drugs& Cosmetics Act 1940 and Rules 1945, amended 11.03.2020 is stored at ILBS and will be used in this trial.

The tests for Donors:

1. Real-time PCR for SARS-CoV-2: Nasal swab samples will be taken prior to donation and tested for SARS-CoV-2 by real-time PCR method it the donor does not have two negative reports 24 hrs apart.

Antibody Titers of Convalescent Plasma and Patients Plasma by ELISA

For Donors:

The titre of serum neutralizing antibody which is the spike protein antibody, directed against the SARS-CoV-2 RBD (receptor binding domain) proteins. The titre will be done by IgG ELISA or by Rapid IgG antibody titre. The minimum titre of 80 is needed for the use of convalescent in patients.

For recipients:

1. Real-time PCR for SARS-CoV-2:

   Nasal swab samples will be taken prior to transfusion and tested for SARS-CoV-2 by real-time PCR method. The test should be positive for eligibility of the recipient along with clinical criteria for COVID-19.
2. Antibody titre: The serum of each recipient will be obtained and IgG antibody titre by enzyme-linked immune-sorbent assay (ELISA) or Rapid IgG antibody method will be tested one day prior to the convalescent plasma transfusion. Changes of IgG antibody titre before and after convalescent plasma transfusion in patients will be studied. The serum will be stored for neutralizing antibody titers by plaque reduction will be done subject to availability.

Study Population:

Adult patients with severe COVID -19 infections defined as WHO Interim Guidance and the Guideline of Diagnosis and Treatment of COVID-19 of National Health Commission of China (version 5.0) with confirmation by real-time RT-PCR assay with severe disease i.e. meeting any 2 of the following criteria

1. Patients on ventilator (in last 24 hours)
2. Respiratory distress, RR ≥30 beats/min
3. Oxygen saturation level less than 90% in resting state
4. Partial pressure of oxygen (PaO2)/oxygen concentration (FiO2) ≤ 300 mmHg
5. Lung infiltrates > 50% within 24 to 48 hours

Study Design:

An open label randomized controlled trial. The study group will comprise of 400 adult patients with severe COVID -19 as detailed above.

Randomization will be done in the ratio of 1:1 in with 200 patients in the treatment arm and 200 patients in the control arm. Allocation concealment will be done by Sequentially Numbered Opaque Sealed Envelopes (SNOSE) method.

Intervention Arm: Two doses of 250 ml Convalescent plasma from recovered COVID-19 patients + Standard of Care will be given to severely sick COVID-19 patients in the treatment arm Control Arm: Standard of Care will be given to severely sick COVID-19 patients in the control arm Details of Standard of Care The Ministry of Health and Family Welfare has issued detailed guidelines for the management of sCOVID-19 based on varying grades of severity which may be periodically updated. For the management of ARDS or sepsis the respective guidelines issued by ARDSNet and Surviving Sepsis campaign will be followed. Other institutional protocols for supportive management will be implemented. (Ref: Guidelines on Clinical Management of COVID-19. MoHFW, GoI.2020.) Monitoring and Assessment: Daily until clinical improvement Adverse Effects: Will be documented Stopping rule: None (C) The expected outcome of the project: Investigator expect convalescent plasma therapy to be a safe and efficacious therapy based on our pilot RCT. This study will determine if there is a clinical improvement /mortality benefit and further elaborate on its safety in patients with severe COVID-19

ELIGIBILITY:
Recipient Inclusion Criteria:

- Patients with severe COVID-19 will be considered for randomization and will be transfused convalescent plasma within 3 days of symptom onset (Severe COVID-19) Severe COVID -19 defined by WHO Interim Guidance and the Guideline of Diagnosis and Treatment of COVID-19 of National Health Commission of China (version 5.0) along with confirmation by real-time RT-PCR assay with severe disease i.e. meeting any 2 of the following criteria-

* Patients on ventilator (in last 24 hours)
* Respiratory distress, RR ≥30 beats/min
* Oxygen saturation level less than 90 % in resting state
* Partial pressure of oxygen (PaO2)/oxygen concentration (FiO2) ≤ 300 mmHg
* Lung infiltrates > 50% within 24 to 48 hours

Recipient Exclusion Criteria:

* Patient/ family members who do not give consent to participate in the study.
* Patients with age less than 18 years
* Patients presenting with multi-organ failure
* Pregnancy
* Individuals with HIV and Viral Hepatitis and Cancer
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Hemodynamic instability requiring vasopressors
* Previous history of allergy to plasma
* Cirrhosis
* Severe renal impairment with GFR< 30ml/min or recipients of RRT, peritoneal dialysis
* Patients with uncontrolled diabetes mellitus, hypertension, arrhythmias and unstable Angina

Donor Inclusion Criteria for Plasmapheresis

* Virologically documented (PCR positive by nasopharyngeal swab) who is recovered and free of symptoms for 14 days.
* Has tested negative for SARS CoV 2 on two consecutive tests 24 hrs apart.
* Fulfill all criteria of donor eligibility for donor Plasmapheresis under the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020
* Females who have been pregnant may be tested for anti-HLA antibodies and eligible if negative for the same.

Donors Exclusion Criteria:

* Do not fulfill all criteria of donor eligibility for donor Plasmapheresis under
* the Drugs & Cosmetics Act 1940 and Rules 1945, amended 11.03.2020
* Females who have been pregnant and have not been tested for HLA antibodies or are HLA antibody positive if tested and previously transfused donors (to prevent TRALI)
* Donors who have taken steroids during treatment for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of convalescent plasma in severe COVID 19 patients in time to clinical improvement (Clinical improvement: Reduction of two points in ordinal scale or live discharge from the intensive care unit, whichever is earlier) | Day 28
  The six-point scale is as follows:
  1. death=6;
  2. hospital admission for extracorporeal membrane oxygenation or mechanical ventilation=5;
  3. hospital admission for non-invasive ventilation or high-flow oxygen therapy=4;
  4. hospital admission for oxygen therapy (but not requiring high-flow or non-invasive ventilation)=3;
  5. hospital admission but not requiring oxygen therapy=2;
  6. discharged or having reached discharge criteria (defined as clinical recovery-ie, normalization of pyrexia, respiratory rate 94% on room air, and relief of cough, all maintained for at least 72 h)=1.

SECONDARY OUTCOMES:
Proportion of patients in each category according to the ordinal scale | 48 hours
Proportion of patients in each category according to the ordinal scale | 7 day
Proportion of patients in each category according to the ordinal scale | Day 14
Proportion of patients in each category according to the ordinal scale | Day 28
Duration of oxygen therapy in both groups | Day 28
Duration of hospital stay in both groups | Day 28
Proportion of patients on mechanical ventilation at day 7 in both groups | Day 7
Mortality in both groups | Day 7
Mortality in both groups | Day 28
Duration of Intensive Care Unit stay | Day 28
Incidence of adverse effects in both groups | Day 28
Presence of antibodies against SARS-CoV-2 in serum after plasma administration | Day 0
  IgG Titres against S1, RBD antigen, and SARS CoV2 neutralizing antibody titres
Presence of antibodies against SARS-CoV-2 in serum after plasma administration | Day 3
  IgG Titres against S1, RBD antigen, and SARS CoV2 neutralizing antibody titres
Presence of antibodies against SARS-CoV-2 in serum after plasma administration | Day 7
  IgG Titres against S1, RBD antigen, and SARS CoV2 neutralizing antibody titres
Presence of antibodies against SARS-CoV-2 in serum after plasma administration | Day 14
  IgG Titres against S1, RBD antigen, and SARS CoV2 neutralizing antibody titres
Change in Cytokines in both groups | Day 28
Change in acute phase reactants in both groups | Day 28
  Serum ferritin
Correlation of the titers in COVID-19 convalescent plasma donors with duration of illness, the severity of symptoms, duration of hospital stay, drugs used in therapy, duration between recovery, and donation. | Day 28

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi
  - Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Super Speciality Hospital, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication till 5 years
Access Criteria: It will be available for researcher scientist & government agencies.

REFERENCES:
- [Derived] Bajpai M, Maheshwari A, Dogra V, Kumar S, Gupta E, Kale P, Saluja V, Thomas SS, Trehanpati N, Bihari C, Agarwal R, Bharti P, Shankar P, Hussain J, Chhabra K, Gupta A, Narayanan A, Agarwal S, Jain S, Bhardwaj A, Kumar G, Yadav BK, Sarin SK. Efficacy of convalescent plasma therapy in the patient with COVID-19: a randomised control trial (COPLA-II trial). BMJ Open. 2022 Apr 6;12(4):e055189. doi: 10.1136/bmjopen-2021-055189. PMID 35387813